CLINICAL TRIAL: NCT02641418
Title: Optimising the Efficacy, Patient Perception and Uptake of an Exercise Programme in People in Intermittent Claudication
Acronym: SEIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hull University Teaching Hospitals NHS Trust (Other Government)
Collaborators: University of Hull (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: R1808
Record Dates: First submitted 2015-08-25; First posted 2015-12-29 (Estimated); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Vascular Disease; Intermittent Claudication
Keywords: Exercise
MeSH Terms: conditions — Vascular Diseases; Intermittent Claudication; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Exercise (Other): only 1 arm to trial
  Interventions: Other: Supervised exercise programme

INTERVENTIONS:
Other: Supervised exercise programme — supervised exercise programme

SUMMARY:
Background: Peripheral arterial disease is a result of atherosclerotic occlusion in the major arteries supplying the lower limbs and is associated with an increased risk of mortality and morbidity. It results in restricted blood flow to the skeletal muscles causing intermittent claudication (IC). IC presents as cramp like pain affecting 5% of the population >50 years and is associated with a substantial reduction in walking capacity, quality of life and diminished physical function. Supervised exercise programmes have been demonstrated to improve maximum walking distances and NICE recommends group-based supervised exercise for treating patients with IC. However, there is significant variability in the impact of treatment across studies and little agreement on the underlying mechanism whereby exercise increases functional outcomes. Potential mechanisms include skeletal muscle metabolism, VO2 max, anaerobic threshold and endothelial function. Studies are needed to better understand how exercise improves outcome and in whom, so as to better refine and target the treatment.

The participation of patients with IC in exercise programmes is low. The investigators need to understand factors influencing participation so that we can improve the number of patients with IC benefiting from the programme

The research consists of two workstreams:

Workstream one

Objective:

Assess the extent to which patient baseline characteristics and candidate physiological mechanisms are associated with clinical improvement in IC patients participating in an exercise programme

Patients: Patients with documented IC referred from a Vascular Consultant. Eligible patients will be invited to participate in a 12 week supervised exercise programme.

Testing Schedule: Measurements will be recorded at baseline (prior to exercise), immediately after the completion of the exercise programme and then three months after. Measurements include:

Baseline characteristics that might predict outcome:

* Quality of life using the VascuQol questionnaire
* Clinical indicators of lower limb function: Ankle brachial pressure index (ABPI), intermittent claudication distance (ICD), Maximum walking distance (MWD).

Candidate physiological mechanisms

* Aerobic capacity (VO2 max & AT)
* Muscular strength and endurance
* Muscle morphology (including muscle thickness, pennation angle, fascicle length and elastography)
* Endothelial function (sheer stress response as measured by flow mediated dilation)

Analysis: Regression analysis will be used to explain variation in patient maximum walking distance at 3 months. The regression will use 9 candidate measures of physiological response and 3 baseline measures to explore what mechanism and patient factors may be associated with clinical improvements. 100 patients recruited over 2 years will give a 90% power to detect an additional increase in variability in MWD explained by each candidate measure of around 5% at the a 0.05 significance level.

This research will be used to identify which types of exercise may be most influential in improving outcome and in which patients.

Workstream two

Objective:

Explore the reasons behind patients' participation, non-participation in, experience of and adherence to the exercise programme.

Study Design: An interview study of patients with IC routinely referred for supervised exercise. Three groups of patients will be invited to participate. Those who:

* Choose not to participate in the exercise programme (Group A)
* Agree to participate in the exercise programme (Group B).
* Agree to participate but discontinue after at least one session (Group C).

Semi-structured face-to-face interviews with 20 patients per group, interviews will be conducted using a topic guide to ensure consistency. The format will be flexible to allow participants to generate naturalistic data on what they consider as important and / or successful in terms of outcome. Data will be analysed thematically and managed using Nvivo software - the approach will be inductive and iterative.

This research will be used to redesign the current exercise programme to improve participation and so the impact of exercise in patients with IC.

ELIGIBILITY:
Inclusion Criteria:

* Patients with IC not referred for surgery
* Community dwelling adults aged forty five or over
* Ankle brachial index ABPI less than 0.9 at rest or a drop of more than 20 after exercise testing
* Ability to walk unaided
* English speaking and able to understand simple protocol instructions

Exclusion Criteria:

* Participants who are unable to provide informed consent
* Severe cardiovascular, musculo-skeletal or pulmonary illness precluding participation in the supervised exercise
* Critical limb ischaemia
* Active treatment for cancer

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2015-05; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Patient maximum walking distance | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Hull Royal Infirmary, Hull, East Riding Of Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Harwood AE, Totty JP, Pymer S, Huang C, Hitchman L, Carradice D, Wallace T, Smith GE, Chetter IC. Cardiovascular and musculoskeletal response to supervised exercise in patients with intermittent claudication. J Vasc Surg. 2019 Jun;69(6):1899-1908.e1. doi: 10.1016/j.jvs.2018.10.065. Epub 2018 Dec 21. PMID 30583899
- See also: Cardiovascular and musculoskeletal response to supervised exercise in patients with intermittent claudication. — https://www.ncbi.nlm.nih.gov/pubmed/30583899